CLINICAL TRIAL: NCT03871491
Title: Prevention of Maternal and Neonatal Death/Infections With a Single Oral Dose of Azithromycin in Women in Labor (in Low- and Middle-income Countries): a Randomized Controlled Trial
Brief Title: Azithromycin-Prevention in Labor Use Study (A-PLUS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NICHD Global Network for Women's and Children's Health (Network)
Collaborators: University of Alabama at Birmingham (Other); University Teaching Hospital, Lusaka, Zambia (Other); University of North Carolina, Chapel Hill (Other); Kinshasa School of Public Health (Other); University of Colorado, Denver (Other); Institute of Nutrition of Central America and Panama (Other); University of Virginia (Other); International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Thomas Jefferson University (Other); Columbia University (Other); Aga Khan University (Other); Boston University (Other); Lata Medical Research Foundation, Nagpur (Other); Indiana University School of Medicine (Other); Moi Univeristy (Other); RTI International (Other); Bill and Melinda Gates Foundation (Other); Jawaharlal Nehru Medical College (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CP Azithromycin; U24HD092094 (NIH)
Record Dates: First submitted 2019-03-05; First posted 2019-03-12 (Actual); Results first posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Maternal Death; Maternal Infections Affecting Fetus or Newborn; Neonatal SEPSIS; Maternal Sepsis During Labor; Neonatal Death; Postpartum Sepsis
Keywords: maternal sepsis; maternal death; neonatal sepsis; neonatal death; azithromycin; Democratic Republic of Congo; Zambia; Guatemala; Bangladesh; India; Pakistan; Kenya; COVID-19
MeSH Terms: conditions — Maternal Death; Neonatal Sepsis; Perinatal Death; Puerperal Infection; Pregnancy Complications, Infectious; COVID-19 | interventions — Azithromycin

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, parallel multicenter clinical trial. Women in labor will be randomized with one-to-one ratio to intervention/placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Both the azithromycin and placebo will be procured from the same manufacturer. The packaging will be standardized across sites and will be labeled as: "Azithromycin 2 g or Placebo", with the expiration data and a unique identifier.
  Clinical and research staff as well as the women will be masked to treatment status unless there is a serious adverse event potentially related to the treatment modality that requires unmasking for safety reasons. There will be one pharmacist at each site who will monitor randomization, drug supply, and safety. If concerns about randomization or participant safety are identified, the data coordinating center will authorize and instruct the study pharmacist to apply un-masking procedures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The study intervention is a single 2 g dose of directly observed oral azithromycin.
  Interventions: Drug: Azithromycin
- Placebo (Placebo Comparator): By random allocation, participants will receive four oral placebo pills containing a non-antimicrobial agent directly after randomization.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin — The study intervention is a single 2 g dose of directly observed oral azithromycin, to be administered as four 500 mg pills or tablets directly after randomization. By random allocation, participants will receive 2 g of oral azithromycin.
  Arms: Intervention
Drug: Placebo — Identical appearing placebo, administered as a single oral dose directly after randomization.
  Arms: Placebo

SUMMARY:
Maternal and neonatal infections are among the most frequent causes of maternal and neonatal deaths, and current antibiotic strategies have not been effective in preventing many of these deaths. Recently, a randomized clinical trial conducted in a single site in The Gambia showed that treatment with oral dose of 2 g azithromycin vs. placebo for all women in labor reduced selected maternal and neonatal infections. However, it is unknown if this therapy reduces maternal and neonatal sepsis and mortality. The A-PLUS trial includes two primary hypotheses, a maternal hypothesis and a neonatal hypothesis. First, a single, prophylactic intrapartum oral dose of 2 g azithromycin given to women in labor will reduce maternal death or sepsis. Second, a single, prophylactic intrapartum oral dose of 2 g azithromycin given to women in labor will reduce intrapartum/neonatal death or sepsis.

DETAILED DESCRIPTION:
The A-PLUS Trial is a randomized, placebo-controlled, parallel multicenter clinical trial. The study intervention is a single, prophylactic intrapartum oral dose of 2 g azithromycin, with a comparison with a single intrapartum oral dose of an identical appearing placebo. For the A-PLUS randomized control trial (RCT), a total of 34,000 laboring women from eight research sites in sub-Saharan Africa, South Asia, and Latin America will be randomized with one-to-one ratio to intervention/placebo. In response to the global coronavirus pandemic, research sites will also collect data on COVID-19 signs/symptoms, diagnosis, and treatment in order to estimate the incidence of infection and evaluate the impact of the pandemic on the target population.

Prior to the initiation of the A-PLUS RCT, research sites will conduct an observational pilot study using the RCT's planned infrastructure in order to characterize the current practices at participating research facilities and optimize the identification of suspected infection for the RCT. The information obtained in the pilot study will be used to validate estimates of intrapartum deaths, maternal sepsis, and neonatal sepsis used in the sample size calculations for the RCT. Finally, the pilot study will allow the research sites to inventory and upgrade local capacity to conduct routine cultures during the RCT.

A maximum of 16,000 women, separate from the sample for the main trial, will be enrolled in the pilot, across all eight research sites, with no more than 2000 women enrolled at any individual site. Research sites will be eligible to transition to the RCT when a minimum of 600 participants have been enrolled in the pilot study with evidence of (a) high rates of follow-up; (2) acceptable data quality and completeness; and (3) there are no concerns about identification and reporting of infection.

Given the clinical benefits of intrapartum azithromycin so far reported in two trials and the likelihood that it may become the usual practice if the investigator's large RCT confirms the reported benefits, it is important to monitor antibiotic resistance to determine the safety of azithromycin prophylaxis. Therefore, the RCT will also include an ancillary study (referred to as the antimicrobial resistance (AMR) sub-study) to monitor antimicrobial resistance and maternal and newborn microbiome effects of the single dose of prophylactic azithromycin using the following methodology

1. For all mothers enrolled in the RCT and their infants:

   a. Routine clinical monitoring at baseline and three post-partum time points (3 days, 7 days, and 42 days), with culture and sensitivity testing in cases of suspected bacterial infections;
2. Among a subset of 1000 randomly selected maternal-infant dyads:

   1. Serial susceptibility monitoring of antimicrobial resistance patterns (including azithromycin resistance) from selected maternal and newborn flora through culture and sensitivity testing. Serial monitoring will be conducted at baseline and three post-partum time points (1 week, 6 weeks, and 3 months).
   2. Serial microbiome collection and storage of specimens for future testing to monitor maternal and newborn microbiome status of selected sites.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in labor ≥28 weeks Gestational Age (GA) (by best estimate) with a pregnancy with one or more live fetuses who plan to deliver vaginally in a facility.
* Admitted to health facility with clear plan for spontaneous or induced delivery.
* Live fetus must be confirmed via a fetal heart rate by Doptone prior to randomization.
* ≥18 years of age or minors 14-17 years of age in countries where married or pregnant minors (or their authorized representatives) are legally permitted to give consent.
* Have provided written informed consent.
* Pregnant women in labor ≥28 weeks GA (by best estimate) with a pregnancy with one or more live fetuses who plan to deliver vaginally in a facility.
* Admitted to health facility with clear plan for spontaneous or induced delivery.
* Live fetus must be confirmed via presence of a fetal heart rate prior to randomization.
* ≥18 years of age or minors 14-17 years of age in countries where married or pregnant minors (or their authorized representatives) are legally permitted to give consent.
* Have provided written informed consent [Note: written informed consent may be obtained during antenatal care, but verbal re-confirmation may be needed (per local regulations) at the time of randomization].

Exclusion Criteria:

* Non-emancipated minors (as per local regulations)
* Evidence of chorioamnionitis or other infection requiring antibiotic therapy at time of eligibility (however, women given single prophylactic antibiotics with no plans to continue after delivery should not be excluded).
* Arrhythmia or known history of cardiomyopathy.
* Allergy to azithromycin or other macrolides that is self-reported or documented in the medical record.
* Any use of azithromycin, erythromycin, or other macrolide in the 3 days or less prior to randomization.
* Plan for cesarean delivery prior to randomization.
* Preterm labor undergoing management with no immediate plan to proceed to delivery.
* Advanced stage of labor (>6 cm or 10 cm cervical dilation per local standards) and pushing or too distressed to understand, confirm, or give informed consent regardless of cervical dilation.
* Are not capable of giving consent due to other health problems such as obstetric emergencies (for example, antepartum hemorrhage) or mental disorder.
* Any other medical conditions that may be considered a contraindication per the judgment of the site investigator.
* Previous randomization in the trial.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58747 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marion Koso-Thomas, MD, Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (8):
- ICDDRB, Dhaka, Bangladesh
- Kinshasa School of Public Health, Kinshasa, Democratic Republic of the Congo
- Institute for Nutrition of Central America and Panama (INCAP), Guatemala City, Guatemala
- India (2):
  - Jawaharlal Nehru Medical College, Belagām
  - Lata Medical Research Foundation, Nagpur
- Moi University School of Medicine, Eldoret, Kenya
- The Aga Khan University, Karachi, Pakistan
- University Teaching Hospital, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data will be made available through the NICHD Data and Specimen Hub (N-DASH) system, a publicly accessible online archive, following publication of the primary paper.
Supporting Information: Study Protocol, SAP
Time Frame: No more than one year after publication of the primary paper. No end date.
Access Criteria: Deidentified participant data will be made available through the NICHD Data and Specimen Hub (N-DASH) system, a publicly accessible online archive. Investigators interested in data and access are required to submit their request through N-DASH, per the requirements of the DASH policy. This includes a brief description of the proposed use of the research data, a signed NICHD DASH Data Use Agreement, and IRB approval, exemption, or declaration that the research does not involve human subjects.
URL: https://dash.nichd.nih.gov/resource/policies

REFERENCES:
- [Background] WHO Recommendations for Prevention and Treatment of Maternal Peripartum Infections. Geneva: World Health Organization; 2015. Available from http://www.ncbi.nlm.nih.gov/books/NBK327079/ PMID 26598777
- [Background] Liu L, Oza S, Hogan D, Perin J, Rudan I, Lawn JE, Cousens S, Mathers C, Black RE. Global, regional, and national causes of child mortality in 2000-13, with projections to inform post-2015 priorities: an updated systematic analysis. Lancet. 2015 Jan 31;385(9966):430-40. doi: 10.1016/S0140-6736(14)61698-6. Epub 2014 Sep 30. PMID 25280870
- [Background] African Neonatal Sepsis Trial (AFRINEST) group; Tshefu A, Lokangaka A, Ngaima S, Engmann C, Esamai F, Gisore P, Ayede AI, Falade AG, Adejuyigbe EA, Anyabolu CH, Wammanda RD, Ejembi CL, Ogala WN, Gram L, Cousens S. Simplified antibiotic regimens compared with injectable procaine benzylpenicillin plus gentamicin for treatment of neonates and young infants with clinical signs of possible serious bacterial infection when referral is not possible: a randomised, open-label, equivalence trial. Lancet. 2015 May 2;385(9979):1767-1776. doi: 10.1016/S0140-6736(14)62284-4. Epub 2015 Apr 1. PMID 25842221
- [Background] Baqui AH, Saha SK, Ahmed AS, Shahidullah M, Quasem I, Roth DE, Samsuzzaman AK, Ahmed W, Tabib SM, Mitra DK, Begum N, Islam M, Mahmud A, Rahman MH, Moin MI, Mullany LC, Cousens S, El Arifeen S, Wall S, Brandes N, Santosham M, Black RE; Projahnmo Study Group in Bangladesh. Safety and efficacy of alternative antibiotic regimens compared with 7 day injectable procaine benzylpenicillin and gentamicin for outpatient treatment of neonates and young infants with clinical signs of severe infection when referral is not possible: a randomised, open-label, equivalence trial. Lancet Glob Health. 2015 May;3(5):e279-87. doi: 10.1016/S2214-109X(14)70347-X. Epub 2015 Apr 1. PMID 25841891
- [Background] Mir F, Nisar I, Tikmani SS, Baloch B, Shakoor S, Jehan F, Ahmed I, Cousens S, Zaidi AK. Simplified antibiotic regimens for treatment of clinical severe infection in the outpatient setting when referral is not possible for young infants in Pakistan (Simplified Antibiotic Therapy Trial [SATT]): a randomised, open-label, equivalence trial. Lancet Glob Health. 2017 Feb;5(2):e177-e185. doi: 10.1016/S2214-109X(16)30335-7. Epub 2016 Dec 15. PMID 27988146
- [Background] Zaidi AK, Tikmani SS, Sultana S, Baloch B, Kazi M, Rehman H, Karimi K, Jehan F, Ahmed I, Cousens S. Simplified antibiotic regimens for the management of clinically diagnosed severe infections in newborns and young infants in first-level facilities in Karachi, Pakistan: study design for an outpatient randomized controlled equivalence trial. Pediatr Infect Dis J. 2013 Sep;32 Suppl 1(Suppl 1 Innovative Treatment Regimens for Severe Infections in Young Infants):S19-25. doi: 10.1097/INF.0b013e31829ff7aa. PMID 23945571
- [Background] Gibbs RS. Clinical risk factors for puerperal infection. Obstet Gynecol. 1980 May;55(5 Suppl):178S-184S. doi: 10.1097/00006250-198003001-00045. PMID 6990333
- [Background] World Health Organization. (2015). WHO Statement on Caesarean Section Rates. Retrieved August 22, 2018, from http://www.who.int/reproductivehealth/publications/maternal_perinatal_health/cs-statement/en/
- [Background] Mackeen AD, Packard RE, Ota E, Berghella V, Baxter JK. Timing of intravenous prophylactic antibiotics for preventing postpartum infectious morbidity in women undergoing cesarean delivery. Cochrane Database Syst Rev. 2014 Dec 5;2014(12):CD009516. doi: 10.1002/14651858.CD009516.pub2. PMID 25479008
- [Background] Smaill FM, Grivell RM. Antibiotic prophylaxis versus no prophylaxis for preventing infection after cesarean section. Cochrane Database Syst Rev. 2014 Oct 28;2014(10):CD007482. doi: 10.1002/14651858.CD007482.pub3. PMID 25350672
- [Background] Gyte GM, Dou L, Vazquez JC. Different classes of antibiotics given to women routinely for preventing infection at caesarean section. Cochrane Database Syst Rev. 2014 Nov 17;2014(11):CD008726. doi: 10.1002/14651858.CD008726.pub2. PMID 25402227
- [Background] Tita ATN, Rouse DJ, Blackwell S, Saade GR, Spong CY, Andrews WW. Emerging concepts in antibiotic prophylaxis for cesarean delivery: a systematic review. Obstet Gynecol. 2009 Mar;113(3):675-682. doi: 10.1097/AOG.0b013e318197c3b6. PMID 19300334
- [Background] Tita AT, Szychowski JM, Boggess K, Saade G, Longo S, Clark E, Esplin S, Cleary K, Wapner R, Letson K, Owens M, Abramovici A, Ambalavanan N, Cutter G, Andrews W; C/SOAP Trial Consortium. Adjunctive Azithromycin Prophylaxis for Cesarean Delivery. N Engl J Med. 2016 Sep 29;375(13):1231-41. doi: 10.1056/NEJMoa1602044. PMID 27682034
- [Background] Oluwalana C, Camara B, Bottomley C, Goodier S, Bojang A, Kampmann B, Ceesay S, D'Alessandro U, Roca A. Azithromycin in Labor Lowers Clinical Infections in Mothers and Newborns: A Double-Blind Trial. Pediatrics. 2017 Feb;139(2):e20162281. doi: 10.1542/peds.2016-2281. PMID 28130432
- [Background] World Health Organization. (2017). Statement on maternal sepsis. Retrieved Ausust 22, 2018, from http://www.who.int/reproductivehealth/publications/maternal_perinatal_health/maternalsepsis-statement/en/
- [Background] Reinhart K, Daniels R, Kissoon N, Machado FR, Schachter RD, Finfer S. Recognizing Sepsis as a Global Health Priority - A WHO Resolution. N Engl J Med. 2017 Aug 3;377(5):414-417. doi: 10.1056/NEJMp1707170. Epub 2017 Jun 28. No abstract available. PMID 28658587
- [Background] van Dillen J, Zwart J, Schutte J, van Roosmalen J. Maternal sepsis: epidemiology, etiology and outcome. Curr Opin Infect Dis. 2010 Jun;23(3):249-54. doi: 10.1097/QCO.0b013e328339257c. PMID 20375891
- [Background] Roca A, Oluwalana C, Bojang A, Camara B, Kampmann B, Bailey R, Demba A, Bottomley C, D'Alessandro U. Oral azithromycin given during labour decreases bacterial carriage in the mothers and their offspring: a double-blind randomized trial. Clin Microbiol Infect. 2016 Jun;22(6):565.e1-9. doi: 10.1016/j.cmi.2016.03.005. Epub 2016 Mar 26. PMID 27026482
- [Background] Harper LM, Kilgore M, Szychowski JM, Andrews WW, Tita ATN. Economic Evaluation of Adjunctive Azithromycin Prophylaxis for Cesarean Delivery. Obstet Gynecol. 2017 Aug;130(2):328-334. doi: 10.1097/AOG.0000000000002129. PMID 28697108
- [Background] Andrews WW, Hauth JC, Cliver SP, Savage K, Goldenberg RL. Randomized clinical trial of extended spectrum antibiotic prophylaxis with coverage for Ureaplasma urealyticum to reduce post-cesarean delivery endometritis. Obstet Gynecol. 2003 Jun;101(6):1183-9. doi: 10.1016/s0029-7844(03)00016-4. PMID 12798523
- [Background] Tita AT, Hauth JC, Grimes A, Owen J, Stamm AM, Andrews WW. Decreasing incidence of postcesarean endometritis with extended-spectrum antibiotic prophylaxis. Obstet Gynecol. 2008 Jan;111(1):51-6. doi: 10.1097/01.AOG.0000295868.43851.39. PMID 18165392
- [Background] Tita AT, Owen J, Stamm AM, Grimes A, Hauth JC, Andrews WW. Impact of extended-spectrum antibiotic prophylaxis on incidence of postcesarean surgical wound infection. Am J Obstet Gynecol. 2008 Sep;199(3):303.e1-3. doi: 10.1016/j.ajog.2008.06.068. PMID 18771992
- [Background] Watts DH, Eschenbach DA, Kenny GE. Early postpartum endometritis: the role of bacteria, genital mycoplasmas, and Chlamydia trachomatis. Obstet Gynecol. 1989 Jan;73(1):52-60. PMID 2783262
- [Background] Hoyme UB, Kiviat N, Eschenbach DA. Microbiology and treatment of late postpartum endometritis. Obstet Gynecol. 1986 Aug;68(2):226-32. PMID 3737039
- [Background] Emmons SL, Krohn M, Jackson M, Eschenbach DA. Development of wound infections among women undergoing cesarean section. Obstet Gynecol. 1988 Oct;72(4):559-64. PMID 3419735
- [Background] Roberts S, Maccato M, Faro S, Pinell P. The microbiology of post-cesarean wound morbidity. Obstet Gynecol. 1993 Mar;81(3):383-6. PMID 8437791
- [Background] Rosene K, Eschenbach DA, Tompkins LS, Kenny GE, Watkins H. Polymicrobial early postpartum endometritis with facultative and anaerobic bacteria, genital mycoplasmas, and Chlamydia trachomatis: treatment with piperacillin or cefoxitin. J Infect Dis. 1986 Jun;153(6):1028-37. doi: 10.1093/infdis/153.6.1028. PMID 3701114
- [Background] Andrews WW, Shah SR, Goldenberg RL, Cliver SP, Hauth JC, Cassell GH. Association of post-cesarean delivery endometritis with colonization of the chorioamnion by Ureaplasma urealyticum. Obstet Gynecol. 1995 Apr;85(4):509-14. doi: 10.1016/0029-7844(94)00436-H. PMID 7898825
- [Background] Keski-Nisula L, Kirkinen P, Katila ML, Ollikainen M, Suonio S, Saarikoski S. Amniotic fluid U. urealyticum colonization: significance for maternal peripartal infections at term. Am J Perinatol. 1997 Mar;14(3):151-6. doi: 10.1055/s-2007-994117. PMID 9259918
- [Background] Yoon BH, Romero R, Park JS, Chang JW, Kim YA, Kim JC, Kim KS. Microbial invasion of the amniotic cavity with Ureaplasma urealyticum is associated with a robust host response in fetal, amniotic, and maternal compartments. Am J Obstet Gynecol. 1998 Nov;179(5):1254-60. doi: 10.1016/s0002-9378(98)70142-5. PMID 9822511
- [Background] Ledger WJ. Prophylactic antibiotics in obstetrics-gynecology: a current asset, a future liability? Expert Rev Anti Infect Ther. 2006 Dec;4(6):957-64. doi: 10.1586/14787210.4.6.957. PMID 17181412
- [Background] Guideline: Managing Possible Serious Bacterial Infection in Young Infants When Referral Is Not Feasible. Geneva: World Health Organization; 2015. Available from http://www.ncbi.nlm.nih.gov/books/NBK321136/ PMID 26447263
- [Background] Sutton AL, Acosta EP, Larson KB, Kerstner-Wood CD, Tita AT, Biggio JR. Perinatal pharmacokinetics of azithromycin for cesarean prophylaxis. Am J Obstet Gynecol. 2015 Jun;212(6):812.e1-6. doi: 10.1016/j.ajog.2015.01.015. Epub 2015 Jan 13. PMID 25595580
- [Background] Eberly MD, Eide MB, Thompson JL, Nylund CM. Azithromycin in early infancy and pyloric stenosis. Pediatrics. 2015 Mar;135(3):483-8. doi: 10.1542/peds.2014-2026. PMID 25687145
- [Background] Ray WA, Murray KT, Hall K, Arbogast PG, Stein CM. Azithromycin and the risk of cardiovascular death. N Engl J Med. 2012 May 17;366(20):1881-90. doi: 10.1056/NEJMoa1003833. PMID 22591294
- [Background] Svanstrom H, Pasternak B, Hviid A. Use of azithromycin and death from cardiovascular causes. N Engl J Med. 2013 May 2;368(18):1704-12. doi: 10.1056/NEJMoa1300799. PMID 23635050
- [Background] Hoffman MK, Goudar SS, Kodkany BS, Goco N, Koso-Thomas M, Miodovnik M, McClure EM, Wallace DD, Hemingway-Foday JJ, Tshefu A, Lokangaka A, Bose CL, Chomba E, Mwenechanya M, Carlo WA, Garces A, Krebs NF, Hambidge KM, Saleem S, Goldenberg RL, Patel A, Hibberd PL, Esamai F, Liechty EA, Silver R, Derman RJ. A description of the methods of the aspirin supplementation for pregnancy indicated risk reduction in nulliparas (ASPIRIN) study. BMC Pregnancy Childbirth. 2017 May 3;17(1):135. doi: 10.1186/s12884-017-1312-x. PMID 28468653
- [Background] Goldenberg RL, Saleem S, Ali S, Moore JL, Lokangako A, Tshefu A, Mwenechanya M, Chomba E, Garces A, Figueroa L, Goudar S, Kodkany B, Patel A, Esamai F, Nsyonge P, Harrison MS, Bauserman M, Bose CL, Krebs NF, Hambidge KM, Derman RJ, Hibberd PL, Liechty EA, Wallace DD, Belizan JM, Miodovnik M, Koso-Thomas M, Carlo WA, Jobe AH, McClure EM. Maternal near miss in low-resource areas. Int J Gynaecol Obstet. 2017 Sep;138(3):347-355. doi: 10.1002/ijgo.12219. Epub 2017 Jun 13. PMID 28513837
- [Background] Bonet M, Souza JP, Abalos E, Fawole B, Knight M, Kouanda S, Lumbiganon P, Nabhan A, Nadisauskiene R, Brizuela V, Metin Gulmezoglu A. The global maternal sepsis study and awareness campaign (GLOSS): study protocol. Reprod Health. 2018 Jan 30;15(1):16. doi: 10.1186/s12978-017-0437-8. PMID 29382352
- [Background] Albright CM, Has P, Rouse DJ, Hughes BL. Internal Validation of the Sepsis in Obstetrics Score to Identify Risk of Morbidity From Sepsis in Pregnancy. Obstet Gynecol. 2017 Oct;130(4):747-755. doi: 10.1097/AOG.0000000000002260. PMID 28885400
- [Background] Bowyer L, Robinson HL, Barrett H, Crozier TM, Giles M, Idel I, Lowe S, Lust K, Marnoch CA, Morton MR, Said J, Wong M, Makris A. SOMANZ guidelines for the investigation and management sepsis in pregnancy. Aust N Z J Obstet Gynaecol. 2017 Oct;57(5):540-551. doi: 10.1111/ajo.12646. Epub 2017 Jul 3. PMID 28670748
- [Derived] Sidze L, Moore JL, Carlo WA, Mwenechanya M, Chomba E, Hemingway-Foday JJ, Kavi A, Metgud MC, Goudar SS, Derman R, Lokangaka AL, Tshefu AK, Bauserman MS, Bose CL, Shivkumar P, Waikar M, Patel AB, Hibberd PL, Nyongesa P, Esamai F, Ekhaguere OA, Bucher SL, Jessani S, Tikmani SS, Saleem S, Goldenberg RL, Billah SM, Lennox R, Haque R, Petri WA, Figueroa L, Mazariegos M, Krebs NF, Nolen TL, Koso-Thomas M, McClure EM, Tita ATN; A-PLUS Trial Group. Intrapartum oral azithromycin for maternal infection prophylaxis and the risk of postpartum hemorrhage: A secondary analysis of the A-PLUS trial. Int J Gynaecol Obstet. 2026 Jan 13. doi: 10.1002/ijgo.70777. Online ahead of print. PMID 41527950
- [Derived] Carlo WA, Tita ATN, Moore JL, Mwenechanya M, Chomba E, Hemingway-Foday JJ, Kavi A, Metgud MC, Goudar SS, Derman RJ, Lokangaka A, Tshefu A, Bauserman M, Patterson JK, Shivkumar P, Waikar M, Patel A, Hibberd PL, Nyongesa P, Esamai F, Ekhaguere OA, Bucher S, Jessani S, Tikmani SS, Saleem S, Goldenberg RL, Billah SM, Lennox R, Haque R, Petri W, Mazariegos M, Krebs NF, Babineau DC, McClure EM, Koso-Thomas M; A-PLUS Trial Group. Effectiveness of intrapartum azithromycin to prevent infections in planned vaginal births in low-income and middle-income countries: a post-hoc analysis of data from a multicentre, randomised, double-blind, placebo-controlled trial. Lancet Glob Health. 2025 Apr;13(4):e689-e697. doi: 10.1016/S2214-109X(24)00562-X. PMID 40155106
- [Derived] Patterson JK, Neuwahl S, Kirsch S, Moore JL, Tita ATN, Carlo WA, Lokangaka A, Tshefu A, Mwenechanya M, Chomba E, Kavi A, Metgud MC, Goudar SS, Derman RJ, Shivkumar P, Waikar M, Patel A, Hibberd PL, Nyongesa P, Esamai F, Ekhaguere OA, Bucher S, Jessani S, Tikmani SS, Saleem S, Wylie BJ, Goldenberg RL, Billah SM, Lennox R, Haque R, Petri WA, Mazariegos M, Krebs NF, Hemingway-Foday JJ, Babineau D, Koso-Thomas M, McClure EM, Bauserman M. Cost-effectiveness of intrapartum azithromycin to prevent maternal infection, sepsis, or death in low-income and middle-income countries: a modelling analysis of data from a randomised, multicentre, placebo-controlled trial. Lancet Glob Health. 2025 Apr;13(4):e679-e688. doi: 10.1016/S2214-109X(24)00517-5. PMID 40155105
- [Derived] Hemingway-Foday J, Tita A, Chomba E, Mwenechanya M, Mweemba T, Nolen T, Lokangaka A, Tshefu Kitoto A, Lomendje G, Hibberd PL, Patel A, Das PK, Kurhe K, Goudar SS, Kavi A, Metgud M, Saleem S, Tikmani SS, Esamai F, Nyongesa P, Sagwe A, Figueroa L, Mazariegos M, Billah SM, Haque R, Shahjahan Siraj M, Goldenberg RL, Bauserman M, Bose C, Liechty EA, Ekhaguere OA, Krebs NF, Derman R, Petri WA, Koso-Thomas M, McClure E, Carlo WA. Prevention of maternal and neonatal death/infections with a single oral dose of azithromycin in women in labour in low-income and middle-income countries (A-PLUS): a study protocol for a multinational, randomised placebo-controlled clinical trial. BMJ Open. 2023 Aug 30;13(8):e068487. doi: 10.1136/bmjopen-2022-068487. PMID 37648383
- [Derived] Tita ATN, Carlo WA, McClure EM, Mwenechanya M, Chomba E, Hemingway-Foday JJ, Kavi A, Metgud MC, Goudar SS, Derman R, Lokangaka A, Tshefu A, Bauserman M, Bose C, Shivkumar P, Waikar M, Patel A, Hibberd PL, Nyongesa P, Esamai F, Ekhaguere OA, Bucher S, Jessani S, Tikmani SS, Saleem S, Goldenberg RL, Billah SM, Lennox R, Haque R, Petri W, Figueroa L, Mazariegos M, Krebs NF, Moore JL, Nolen TL, Koso-Thomas M; A-PLUS Trial Group. Azithromycin to Prevent Sepsis or Death in Women Planning a Vaginal Birth. N Engl J Med. 2023 Mar 30;388(13):1161-1170. doi: 10.1056/NEJMoa2212111. Epub 2023 Feb 9. PMID 36757318

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomized, multi-country, double-masked, placebo-controlled trial of azithromycin (single 2g oral dose) initiated during labor, in women who were in labor at 28 weeks' gestation or more and who were planning a vaginal delivery
Pre-assignment Details: Participants were randomly assigned (1:1, stratified by site) to receive azithromycin or placebo tablets of identical appearance, via a sequence generated centrally by the data coordinating center. Mother were randomized and the maternal participant and her baby or babies in the case of multiple pregnancies were enrolled.
Groups:
- Azithromycin Intervention (Mothers): The study intervention is a single 2 g dose of directly observed oral azithromycin.
  Azithromycin: The study intervention is a single 2 g dose of directly observed oral azithromycin, to be administered to maternal participants as four 500 mg pills or tablets directly after randomization which occurs between the onset of labor and delivery. By random allocation, participants will receive 2 g of oral azithromycin.
- Azithromycin Intervention (Neonates): The study intervention is a single 2 g dose of directly observed oral azithromycin.
  Azithromycin: The study intervention is a single 2 g dose of directly observed oral azithromycin, to be administered to maternal participants as four 500 mg pills or tablets directly after randomization which occurs between the onset of labor and delivery. By random allocation, participants will receive 2 g of oral azithromycin. Stillbirths and live births of maternal participants randomized are considered enrolled to the arm which their mother was randomized.
- Placebo (Mothers): By random allocation, participants will receive four oral placebo pills containing a non-antimicrobial agent directly after randomization.
  Placebo: Identical appearing placebo, administered to maternal participants as a single oral dose directly after randomization, which occurs between the onset of labor and delivery.
- Placebo (Neonates): By random allocation, participants will receive four oral placebo pills containing a non-antimicrobial agent directly after randomization.
  Placebo: Identical appearing placebo, administered to maternal participants as a single oral dose directly after randomization, which occurs between the onset of labor and delivery. Stillbirths and live births of maternal participants randomized are considered enrolled to the arm which their mother was randomized.
Period: Overall Study
Arm/Group | Azithromycin Intervention (Mothers) | Azithromycin Intervention (Neonates) | Placebo (Mothers) | Placebo (Neonates)
Started | 14590 | 14687 (14628 neonates and 59 stillbirths) | 14688 | 14782 (14726 neonates and 56 stillbirths)
Treated | 14589 | 14686 (14628 neonates and 59 stillbirths born to women treated) | 14687 | 14781 (14726 neonates and 56 stillbirths born to women treated)
Included in Intention to Treat (ITT) Analysis | 14590 | 14687 (14628 neonates and 59 stillbirths) | 14688 | 14782 (14726 neonates and 59 stillbirths)
Completed | 14526 | 14658 | 14637 | 14756
Not Completed | 64 | 29 | 51 | 26
Not completed — Withdrawal by Subject | 14 | 14 | 14 | 14
Not completed — Physician Decision | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 50 | 15 | 36 | 11

BASELINE CHARACTERISTICS:
Population: Women who were eligible according to the intention-to-treat (ITT) criteria and included in the ITT analysis. Includes baseline data for neonates of randomized maternal participants. Baseline data was not collected for the 115 stillbirths. The number of neonates is larger than the number of maternal participants randomized due to multiple births.
Groups:
- Total: Total of all reporting groups
Arm/Group | Azithromycin Intervention (Mothers) | Azithromycin Intervention (Neonates) | Placebo (Mothers) | Placebo (Neonates) | Total
Number analyzed (Participants) | 14590 | 14687 | 14688 | 14782 | 58747
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Maternal age at enrollment (years) Population: This measure applies to mothers randomized and does not apply to neonates/stillbirths.
  years
    number analyzed (Participants) | 14590 | 0 | 14688 | 0 | 29278
    (all) | 24 [21 to 28] |  | 24 [21 to 28] |  | 24 [21 to 28]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 14590 | 7123 | 14688 | 7190 | 43591
  Male | 0 | 7563 | 0 | 7591 | 15154
  Missing Sex | 0 | 1 | 0 | 1 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Bangladesh | 1406 | 1408 | 1441 | 1446 | 5701
  Pakistan | 1825 | 1841 | 1843 | 1862 | 7371
  Congo, The Democratic Republic of the | 2181 | 2220 | 2192 | 2231 | 8824
  Guatemala | 794 | 794 | 803 | 803 | 3194
  Zambia | 1769 | 1784 | 1765 | 1779 | 7097
  Kenya | 1829 | 1835 | 1844 | 1846 | 7354
  India | 4786 | 4805 | 4800 | 4815 | 19206
Marital status [Count of Participants; unit: Participants] — Population: This measure applies to mothers randomized and does not apply to neonates/stillbirths.
  Participants
    number analyzed (Participants) | 14590 | 0 | 14688 | 0 | 29278
    Married | 13729 |  | 13834 |  | 27563
    Single | 612 |  | 600 |  | 1212
    Other | 248 |  | 253 |  | 501
    Missing | 1 |  | 1 |  | 2
Maternal education [Count of Participants; unit: Participants] — Population: This measure applies to mothers randomized and does not apply to neonates/stillbirths.
  Participants
    number analyzed (Participants) | 14590 | 0 | 14688 | 0 | 29278
    No formal schooling | 3457 |  | 3476 |  | 6933
    1-6 years of schooling | 2002 |  | 2022 |  | 4024
    7-12 years of schooling | 7308 |  | 7325 |  | 14633
    >= 13 years of schooling | 1798 |  | 1842 |  | 3640
    Missing | 25 |  | 23 |  | 48
Primiparous [Count of Participants; unit: Participants] — Primiparous indicates a parity=0. Parity is defined as the number of pregnancies reaching 20 weeks and 0 days of gestation or beyond, regardless of the number of fetuses or outcomes. In cases of multiple pregnancies, parity is only increased with birth of the last fetus. Population: This measure applies to mothers randomized and does not apply to neonates/stillbirths.
  Participants
    number analyzed (Participants) | 14590 | 0 | 14688 | 0 | 29278
    Yes | 6311 |  | 6376 |  | 12687
    No | 8277 |  | 8311 |  | 16588
    Missing | 2 |  | 1 |  | 3
Multiple birth [Count of Participants; unit: Participants] — Multiple birth is the delivery of more than one offspring in a single birth event. For example, twin and triplet deliveries are considered multiple births.
  Participants
    Yes | 99 | 198 | 95 | 190 | 582
    No | 14489 | 14489 | 14592 | 14592 | 58162
    Missing | 2 | 0 | 1 | 0 | 3
Any maternal infection during pregnancy [Count of Participants; unit: Participants] — Maternal infections during pregnancy include group B strep, pneumonia, pyelonephritis, rubella, chlamydia, herpes, syphilis, gonorrhea, HIV, hepatitis B, malaria, urinary tract infection or other infection. Population: This measure applies to mothers randomized and does not apply to neonates/stillbirths.
  Participants
    number analyzed (Participants) | 14590 | 0 | 14688 | 0 | 29278
    Yes | 797 |  | 821 |  | 1618
    No | 13792 |  | 13866 |  | 27658
    Missing | 1 |  | 1 |  | 2
Any maternal condition during pregnancy [Count of Participants; unit: Participants] — Maternal conditions during pregnancy include diabetes, chronic hypertension, hypertensive disorders of pregnancy or other condition. Population: This measure applies to mothers randomized and does not apply to neonates/stillbirths.
  Participants
    number analyzed (Participants) | 14590 | 0 | 14688 | 0 | 29278
    Yes | 1017 |  | 955 |  | 1972
    No | 13572 |  | 13732 |  | 27304
    Missing | 1 |  | 1 |  | 2
Gestational age < 37 weeks [Count of Participants; unit: Participants]
  Yes | 1841 | 1889 | 1895 | 1944 | 7569
  No | 12742 | 12791 | 12789 | 12834 | 51156
  Missing | 7 | 7 | 4 | 4 | 22
Type of labor onset [Count of Participants; unit: Participants] — Population: This measure applies to mothers randomized and does not apply to neonates/stillbirths.
  Participants
    number analyzed (Participants) | 14590 | 0 | 14688 | 0 | 29278
    Induced | 2651 |  | 2724 |  | 5375
    Spontaneous | 11930 |  | 11953 |  | 23883
    Missing | 9 |  | 11 |  | 20
High risk for sepsis before randomization [Count of Participants; unit: Participants] — High risk for sepsis is defined as women who experience prolonged labor (time from labor to randomization >= 18 hours) or prolonged membrane rupture (time from rupture of membranes to randomization >=8 hours). This measure applies to mothers randomized and does not apply to neonates/stillbirths. Population: This measure applies to mothers randomized and does not apply to neonates/stillbirths.
  Participants
    number analyzed (Participants) | 14590 | 0 | 14688 | 0 | 29278
    Yes | 1247 |  | 1283 |  | 2530
    No | 13341 |  | 13404 |  | 26745
    Missing | 2 |  | 1 |  | 3
Prolonged labor >= 18 hours before randomization [Count of Participants; unit: Participants] — Prolonged labor occurs when randomization is 18 or more hours after the onset of labor. Population: This measure applies to mothers randomized and does not apply to neonates/stillbirths.
  Participants
    number analyzed (Participants) | 14590 | 0 | 14688 | 0 | 29278
    Yes | 670 |  | 698 |  | 1368
    No | 13918 |  | 13989 |  | 27907
    Missing | 2 |  | 1 |  | 3
Prolonged rupture of membranes >= 8 hours before randomization [Count of Participants; unit: Participants] — Prolonged rupture of membranes occurs when randomization is 8 or more hours after rupture of membranes. Population: This measure applies to mothers randomized and does not apply to neonates/stillbirths.
  Participants
    number analyzed (Participants) | 14590 | 0 | 14688 | 0 | 29278
    Yes | 615 |  | 632 |  | 1247
    No | 13973 |  | 14055 |  | 28028
    Missing | 2 |  | 1 |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Maternal Death or Sepsis Within 6 Weeks (42 Days) Post-delivery in Intervention vs. Placebo Group.
Description: Maternal death or sepsis within 6 weeks (42 days) post-delivery in intervention vs. placebo group.
Time Frame: Within 6 weeks (42 days)
Population: Intention to treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Placebo
Number analyzed (Participants) | 14,526 | 14,637
Participants | 227 | 344
Statistical Analysis 1: Comparison: Placebo; The null hypothesis is there is no treatment effect on the incidence of maternal death or sepsis within 6 weeks (42 days) post-delivery; Test type: Superiority; p < 0.001, Regression, Logistic — We calculated P values to test each of the primary hypotheses at an alpha level of 0.05 overall, with a nominal alpha level of 0.0001 at the interim analysis; Used multiple imputation for missing outcomes by means of logistic regression imputation; Risk Ratio (RR) = 0.67, 95% CI 2-sided [0.56 to 0.79]

2. Primary Outcome: Intrapartum/Neonatal Death or Sepsis Within 4 Weeks (28 Days) Post-delivery in Intervention vs. Placebo Group
Description: Intrapartum/neonatal death or sepsis within 4 weeks (28 days) post-delivery in intervention vs. placebo group. This outcome is measured among stillbirths and neonates with 28-day status available born to women randomized. The study includes multiple births so there are more stillbirths and neonates than participants enrolled.
Time Frame: Within 4 weeks (28 days) post-delivery
Population: Intention to treat (ITT)
Measure: Count of Participants; unit: Participants
Groups:
- Intervention Arm: The study intervention is a single 2 g dose of directly observed oral azithromycin.
  Azithromycin: The study intervention is a single 2 g dose of directly observed oral azithromycin, to be administered as four 500 mg pills or tablets directly after randomization. By random allocation, participants will receive 2 g of oral azithromycin.
- Placebo Arm: By random allocation, participants will receive four oral placebo pills containing a non-antimicrobial agent directly after randomization.
  Placebo: Identical appearing placebo, administered as a single oral dose directly after randomization.
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 14,658 | 14,756
Participants | 1,540 | 1,526
Statistical Analysis 1: Comparison: Placebo Arm; The null hypothesis is there is no treatment effect on the incidence of Intrapartum/Neonatal Death or Sepsis Within 4 Weeks (28 Days) Post-delivery in Intervention vs. Placebo Group; Test type: Superiority; p = 0.56, Regression, Logistic — [p-value comment as in outcome 1, analysis 1]; Used multiple imputation for missing outcomes by means of logistic regression imputation; Risk Ratio (RR) = 1.02, 95% CI 2-sided [0.95 to 1.09]

3. Secondary Outcome: Maternal Sepsis
Description: Maternal sepsis within 6 weeks (42 days) post-delivery in intervention vs. placebo group.
Time Frame: Within 42 days post-delivery
Population: Intention to treat (ITT). Numbers differ from the participant flow ITT population due to missing data specific to this secondary outcome. Maternal sepsis required a diagnosis of sepsis according to the study algorithm or no diagnosis and follow-up data on/beyond 7 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 14,558 | 14,662
Participants | 219 | 339
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; Risk Ratio (RR) = 0.65, 95% CI 2-sided [0.55 to 0.77]

4. Secondary Outcome: Maternal Death Due to Sepsis
Description: Maternal death due to sepsis using the Global Network algorithm for cause of death
Time Frame: Within 42 days post-delivery
Population: Intention to treat (ITT). Numbers differ from the participant flow ITT population due to missing data specific to this secondary outcome. Maternal death due to sepsis required maternal status at 42-days to be included in the denominator.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 14,526 | 14,635
Participants | 4 | 1
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; Risk Ratio (RR) = 4.04, 95% CI 2-sided [0.45 to 36.14]

5. Secondary Outcome: Chorioamnionitis
Description: Fever (>100.4°F/38°C) in addition to one or more of the following: fetal tachycardia ≥160 bpm, maternal tachycardia >100 bpm, tender uterus between contractions, or purulent/foul smelling discharge from uterus prior to delivery.
Time Frame: Between date/time of randomization and date/time of delivery (up to 120 hours before delivery)
Population: Intention to treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 14,590 | 14,688
Participants | 5 | 8

6. Secondary Outcome: Endometritis
Description: Fever (>100.4°F/38°C) in addition to one or more of maternal tachycardia >100 bpm, tender uterine fundus, or purulent/foul smelling discharge from uterus after delivery.
Time Frame: Within 42 days post-delivery
Population: Intention to treat (ITT). Numbers differ from the participant flow ITT population due to missing data specific to this secondary outcome. Endometritis required a diagnosis according to the study algorithm or no diagnosis and follow-up data on/beyond 7 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 14,558 | 14,659
Participants | 191 | 294
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; Risk Ratio (RR) = 0.66, 95% CI 2-sided [0.55 to 0.79]

7. Secondary Outcome: Cesarean Wound Infection
Description: Wound infection (Purulent infection of a Cesarean wound with or without fever. In the absence of purulence, requires presence of fever >100.4°F/38°C and at least one of the following signs of local infection: pain or tenderness, swelling, heat, or redness around the incision/laceration);
Time Frame: Within 42 days post-delivery
Population: Intention to treat (ITT). This outcome variable is analyzed for the subgroup of women with a cesarean delivery. Numbers differ from the participant flow ITT population due to this subgroup analysis and missing data specific to this secondary outcome. Cesarean wound infection required a diagnosis according to the study algorithm or no diagnosis and follow-up data on/beyond 7 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 2,038 | 2,060
Participants | 77 | 134
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; Risk Ratio (RR) = 0.57, 95% CI 2-sided [0.43 to 0.75]

8. Secondary Outcome: Perineal Wound Infection
Description: Wound infection (Purulent infection of a perineal wound with or without fever. In the absence of purulence, requires presence of fever >100.4°F/38°C and at least one of the following signs of local infection: pain or tenderness, swelling, heat, or redness around the incision/laceration);
Time Frame: Within 42 days post-delivery
Population: Intention to treat (ITT). This outcome variable analyzed for the subgroup of women with a vaginal delivery. Numbers differ from the participant flow ITT population due to this subgroup analysis and missing data specific to this secondary outcome. Perineal wound infection required a diagnosis according to the study algorithm or no diagnosis and follow-up data on/beyond 7 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 12,519 | 12,595
Participants | 149 | 188
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; Risk Ratio (RR) = 0.8, 95% CI 2-sided [0.65 to 0.99]

9. Secondary Outcome: Other Infections
Description: Abdominopelvic abscess (Evidence of pus in the abdomen or pelvis noted during open surgery, interventional aspiration or imaging); Pneumonia (Fever >100.4°F/38°C and clinical symptoms suggestive of lung infection including cough and/or tachypnea >24 breaths/min or radiological confirmation); Pyelonephritis (Fever >100.4°F/38°C and one or more of the following: urinalysis/dip suggestive of infection, costovertebral angle tenderness, or confirmatory urine culture); Mastitis/breast abscess or infection (Fever >100.4°F/38°C and one or more of the following: breast pain, swelling, warmth, redness, or purulent drainage). Other bacterial infection.
Time Frame: Within 42 days post-delivery
Population: Intention to treat (ITT). Numbers differ from the participant flow ITT population due to missing data specific to this secondary outcome. Other infections required a diagnosis according to the study algorithm or no diagnosis and follow-up data on/beyond 7 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 14,558 | 14,657
Participants | 149 | 217
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; Risk Ratio (RR) = 0.69, 95% CI 2-sided [0.56 to 0.85]

10. Secondary Outcome: Use of Subsequent Maternal Antibiotic Therapy
Description: Use of subsequent maternal antibiotic therapy after randomization to 42 days postpartum for any reason.
Time Frame: After randomization to 42 days post-delivery. Randomization occurs between labor onset and delivery (0 to 120 hours before delivery). 42 participants were randomized >120 hours before delivery due to false labor.
Population: Intention to treat (ITT). Numbers differ from the participant flow ITT population due to missing data specific to this secondary outcome. Use of subsequent maternal antibiotic therapy required a yes response or a no response on follow-up data on/beyond 7 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 14,567 | 14,672
Participants | 7,937 | 8,180
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; Risk Ratio (RR) = 0.98, 95% CI 2-sided [0.95 to 1.01]

11. Secondary Outcome: Maternal Initial Hospital Length of Stay
Description: Time from drug administration until initial discharge after delivery (time may vary by site).
Time Frame: Time from drug administration (which occurs between onset of labor and delivery) and discharge from delivery hospital (0 to 45 days)
Population: Intention to treat (ITT). Numbers differ from the participant flow ITT population due to missing data specific to this secondary outcome. Time from drug administration until initial discharge after delivery required non-missing date and time variables for discharge after delivery.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 14,581 | 14,676
days | 1.4 (1.8) | 1.4 (1.9)

12. Secondary Outcome: Maternal Readmissions
Description: Maternal readmissions after delivery discharge and within 42 days of delivery
Time Frame: After delivery discharge and within 42 days post-delivery
Population: Intention to treat (ITT). Numbers differ from the participant flow ITT population due to missing data specific to this secondary outcome. Maternal readmissions required non-missing date of delivery discharge and a readmission or no indication of a readmission and follow-up data on/beyond 7 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 14,552 | 14,646
Participants | 124 | 192
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; Risk Ratio (RR) = 0.65, 95% CI 2-sided [0.52 to 0.82]

13. Secondary Outcome: Maternal Admission to Special Care Units
Description: Maternal admission to special care units
Time Frame: Within 42 days post-delivery (reported during study)
Population: Intention to treat (ITT). Numbers differ from the participant flow ITT population due to missing data specific to this secondary outcome. Maternal admission to special care units required a yes response or a no response on follow-up data on/beyond 7 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 14,560 | 14,662
Participants | 116 | 130
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; Risk Ratio (RR) = 0.90, 95% CI 2-sided [0.70 to 1.15]

14. Secondary Outcome: Maternal Unscheduled Visit for Care
Description: Maternal unscheduled visit for care
Time Frame: Within 42 days post-delivery (reported during study)
Population: Intention to treat (ITT). Numbers differ from the participant flow ITT population due to missing data specific to this secondary outcome. Maternal unscheduled visit for care required a visit for unscheduled care or a no visit reported on follow-up data on/beyond 7 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 14,554 | 14,649
Participants | 1,397 | 1,790
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; Risk Ratio (RR) = 0.79, 95% CI 2-sided [0.73 to 0.84]

15. Secondary Outcome: Maternal GI Symptoms
Description: Maternal GI symptoms including nausea, vomiting, and diarrhea and other reported side effects.
Time Frame: Within 42 days post-delivery (reported during study)
Population: Safety population. This is the Treated row of the participant flow.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 14,589 | 14,687
Participants | 119 | 110
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; Risk Ratio (RR) = 1.09, 95% CI 2-sided [0.84 to 1.41]

16. Secondary Outcome: Neonatal Sepsis
Description: Neonatal sepsis within 4 weeks (28 days) post-delivery in intervention vs. placebo group. This outcome is measured among neonates born to women randomized. The study includes multiple births so there are more neonates than maternal participants enrolled.
Time Frame: Within 28 days post-delivery
Population: Intention to treat (ITT) for live births. Numbers differ from the participant flow ITT population due to missing data specific to this secondary outcome. Neonatal sepsis is defined among live births so excludes stillbirths. Neonatal sepsis required a diagnosis of sepsis according to the study algorithm or no diagnosis and follow-up data on/beyond 7 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 14,570 | 14,652
Participants | 1,433 | 1,407
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.96 to 1.1]

17. Secondary Outcome: Neonatal Death Due to Sepsis
Description: Neonatal death due to sepsis using the Global Network algorithm for causes of death. This outcome is measured among neonates with 28-day status available born to women randomized. The study includes multiple births so there are more neonates than maternal participants enrolled.
Time Frame: Within 28 days post-delivery
Population: Intention to treat (ITT) for live births. Numbers differ from the participant flow ITT population due to missing data specific to this secondary outcome. Neonatal death due to sepsis is defined among live births so excludes stillbirths. Neonatal death due to sepsis required status at 28 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 14,598 | 14,700
Participants | 64 | 62
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; Risk Ratio (RR) = 1.04, 95% CI 2-sided [0.73 to 1.47]

18. Secondary Outcome: Other Neonatal Infections
Description: Other neonatal infections (e.g. eye infection, skin infection). This outcome is measured among neonates born to women randomized. The study includes multiple births so there are more neonates than maternal participants enrolled.
Time Frame: Within 28 days post-delivery
Population: Intention to treat (ITT) for live births. Numbers differ from the participant flow ITT population due to missing data specific to this secondary outcome. Other neonatal infections is defined among live births so excludes stillbirths. Other neonatal infections required a diagnosis according to the study algorithm or no diagnosis and follow-up data on/beyond 7 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 14,573 | 14,657
Participants | 763 | 798
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; Risk Ratio (RR) = 0.97, 95% CI 2-sided [0.88 to 1.07]

19. Secondary Outcome: Neonatal Initial Hospital Length of Stay
Description: Neonatal initial hospital length of stay, defined as time of delivery until initial discharge (time may vary by site). This outcome is measured among neonates born to women randomized. The study includes multiple births so there are more neonates than maternal participants enrolled.
Time Frame: Time from delivery to discharge from delivery hospital (0 to 62 days)
Population: Intention to treat (ITT) for live births. Numbers differ from the participant flow ITT population due to missing data specific to this secondary outcome. Neonatal initial hospital length of stay is defined among live births so excludes stillbirths. Neonatal initial hospital length of stay required non-missing date and time of hospital discharge.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 14,615 | 14,715
days | 1.5 (2.4) | 1.5 (2.1)

20. Secondary Outcome: Neonatal Readmissions
Description: Neonatal readmissions to facility after delivery discharge and within 42 days of delivery. This outcome is measured among neonates born to women randomized. The study includes multiple births so there are more neonates than maternal participants enrolled.
Time Frame: After delivery discharge and within 42 days of delivery
Population: Intention to treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 14,420 | 14,514
Participants | 553 | 518
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; Risk Ratio (RR) = 1.08, 95% CI 2-sided [0.96 to 1.21]

21. Secondary Outcome: Neonatal Admission to Special Care Units
Description: Neonatal admission to special care units. This outcome is measured among neonates born to women randomized. The study includes multiple births so there are more neonates than maternal participants enrolled.
Time Frame: Within 42 days post-delivery (reported during study)
Population: Intention to treat (ITT) for live births. Numbers differ from the participant flow ITT population due to missing data specific to this secondary outcome. Neonatal admission to special care units is defined among live births so excludes stillbirths. Neonatal admission to special care units required a yes response or a no response on follow-up data on/beyond 7 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 14,499 | 14,585
Participants | 951 | 927
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; Risk Ratio (RR) = 1.03, 95% CI 2-sided [0.94 to 1.12]

22. Secondary Outcome: Neonatal Unscheduled Visit for Care
Description: Neonatal unscheduled visit for care. This outcome is measured among neonates born to women randomized. The study includes multiple births so there are more neonates than maternal participants enrolled.
Time Frame: Within 42 days post-delivery (reported during study)
Population: Intention to treat (ITT) for live births. Numbers differ from the participant flow ITT population due to missing data specific to this secondary outcome. Neonatal unscheduled visit for care is defined among live births so excludes stillbirths. Neonatal unscheduled visit for care required a reported unplanned care visit or no unplanned care reported on follow-up data on/beyond 7 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 14,458 | 14,565
Participants | 3,223 | 3,366
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; Risk Ratio (RR) = 0.96, 95% CI 2-sided [0.93 to 1.0]

23. Secondary Outcome: Pyloric Stenosis Within 42 Days of Delivery
Description: Pyloric stenosis within 42 days of delivery, defined as clinical suspicion based on severe vomiting leading to death, surgical intervention (pyloromyotomy) as verified from medical records, or radiological confirmation. This outcome is measured among neonates born to women randomized. The study includes multiple births so there are more neonates than maternal participants enrolled.
Time Frame: Within 42 days post-delivery
Population: Safety population for live births. Numbers differ from Treated in the participant flow because they are live births among treated mothers.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm | Placebo Arm
Number analyzed (Participants) | 14,627 | 14,725
Participants | 8 | 3
Statistical Analysis 1: Comparison: Placebo Arm; Test type: Superiority; Risk Ratio (RR) = 2.68, 95% CI 2-sided [0.71 to 10.1]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored continuously throughout the study from time of randomization (between onset of labor and delivery) through 6-weeks post delivery.
Description: Surveillance of maternal side effects potentially associated with azithromycin was conducted during labor and postpartum. For infants, findings suggestive of pyloric stenosis were assessed during the follow up visits. Maternal and neonatal surveillance included assessment of unintended medical visits and death. Potential side effects with azithromycin use were monitored and reported as a serious adverse event. Adverse events are reported among the Safety population (Treated).
Arm/Group | Azithromycin Intervention (Mothers) | Azithromycin Intervention (Neonates) | Placebo (Mothers) | Placebo (Neonates)
All-Cause Mortality (participants affected / at risk) | 12/14589 | 291/14686 | 11/14687 | 286/14781
Serious Adverse Events (participants affected / at risk) | 3/14589 | 11/14686 | 3/14687 | 8/14781
Other Adverse Events (participants affected / at risk) | 1022/14589 | 8/14686 | 1110/14687 | 3/14781
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Azithromycin Intervention (Mothers) (N=14589) | Azithromycin Intervention (Neonates) (N=14686) | Placebo (Mothers) (N=14687) | Placebo (Neonates) (N=14781)
Maternal death (Pregnancy, puerperium and perinatal conditions) | 3 | 0/0 | 1 | 0/0 — This event applies to mothers only and not neonates (stillbirth or live birth).
Other maternal serious adverse event (Pregnancy, puerperium and perinatal conditions) | 0 | 0/0 | 2 | 0/0 — This event applies to mothers only and not neonates (stillbirth or live birth).
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 0/0 | 1 | 0/0 | 1 — This event applies to neonates only (stillbirth or live birth) and not mothers.
Neonatal death (Pregnancy, puerperium and perinatal conditions) | 0/0 | 9/14627 | 0/0 | 5/14725 — This event applies to neonates only (stillbirth or live birth) and not mothers.
Other neonatal serious adverse event (Pregnancy, puerperium and perinatal conditions) | 0/0 | 1/14627 | 0/0 | 2/14725 — This event applies to neonates only (stillbirth or live birth) and not mothers.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Azithromycin Intervention (Mothers) (N=14589) | Azithromycin Intervention (Neonates) (N=14686) | Placebo (Mothers) (N=14687) | Placebo (Neonates) (N=14781)
Vomited within 15 minutes after study drug administration (Gastrointestinal disorders) | 311 | 0/0 | 279 | 0/0 — This event applies to mothers only and not neonates (stillbirth or live birth).
Feeling faint or dizzy (Cardiac disorders) | 241 | 0/0 | 309 | 0/0 — This event applies to mothers only and not neonates (stillbirth or live birth).
Nausea/vomiting (Gastrointestinal disorders) | 45 | 0/0 | 48 | 0/0 — This event applies to mothers only and not neonates (stillbirth or live birth).
Diarrhea/loose stools (Gastrointestinal disorders) | 76 | 0/0 | 66 | 0/0 — This event applies to mothers only and not neonates (stillbirth or live birth).
Severe abdominal or uterine pain (General disorders) | 170 | 0/0 | 208 | 0/0 — This event applies to mothers only and not neonates (stillbirth or live birth).
Foul-smelling vaginal discharge (General disorders) | 37 | 0/0 | 83 | 0/0 — This event applies to mothers only and not neonates (stillbirth or live birth).
Severe vaginal pain (General disorders) | 309 | 0/0 | 329 | 0/0 — This event applies to mothers only and not neonates (stillbirth or live birth).
GI symptoms and other reported side effects (Gastrointestinal disorders) | 119 | 0/0 | 110 | 0/0 — This event applies to mothers only and not neonates (stillbirth or live birth).
Pyloric stenosis (Gastrointestinal disorders) | 0/0 | 8/14627 | 0/0 | 3/14726 — This event applies to neonates (stillbirth or live birth) and not mothers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-10-13): https://cdn.clinicaltrials.gov/large-docs/91/NCT03871491/Prot_SAP_ICF_000.pdf